CLINICAL TRIAL: NCT04043533
Title: The Effect of an Exercise Program in Reducing the Severity of Postpartum Depression in Women: A Randomized Control Trial
Brief Title: The Effect of an Exercise Program in Reducing the Severity of Postpartum Depression in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Kucukkelepce (Other)
Responsible Party: Sponsor-Investigator, Didem Kucukkelepce, Didem Kucukkelepce, Adiyaman University Research Hospital
Organization: Adiyaman University Research Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AdıyamanUniversty
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with a prospective pretest-posttest experimental design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises Group (Experimental)
  Interventions: Behavioral: Exercises
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Exercises — The women in the experimental group were given information about the benefits of exercises done in the postpartum period, the time to start these exercises, and the exercises to be conducted in three different phases (mild, medium, severe). The first physical exercise practice was done in the FHC together. In line with the recommendations by ACOG (2015), the women were told to do mild and medium level exercises in the first two weeks, at least five days in a week and at least half an hour daily (ACOG, 2015). They were also told that they should do medium and severe level exercises in the following two weeks. They were asked to mark on the form what time, how long, and at what level they did the exercises every day. The education booklet that included this information and the visuals of the exercises were given to the women in the experimental group. In addition, the women were called once a week in order to check whether the training was applied.
  Arms: Exercises Group

SUMMARY:
Aim: This study aims to identify the effectiveness of an exercise program in reducing the severity of postnatal depression in women who had a spontaneous vaginal delivery.

Methods: This randomized control trial was conducted with 65 postpartum women residing in a city located in the south-eastern Turkey. In the first postpartum month, following random assignment of subjects, the experimental group (n=40) performed exercises for four weeks, and the control group (n=40) received standard cares. The participating women were administered the Edinburgh Postpartum Depression Scale.

DETAILED DESCRIPTION:
Postpartum depression is characterized by irritability, guilt, burnout, anxiety, sleep disorders, and somatic symptoms that could have negative effects on the mother, baby, and family.

In a meta-analysis study including 219 prevalence studies from 56 countries that investigated different phases of postpartum using various data collection tools, Hahn-Holbrook et al. (2018) found the depression prevalence at the global level as 17.7% (Hahn-Holbrook, 2018). In Turkey, 23.8% of women in the postpartum period were reported to be suffering from postpartum depression, which underlines the need for health professionals to be concerned about the health of the women in the postpartum period.

Exercises done in the postpartum period are reported to enable psychosocial well-being, less anxiety and depression, better cardiovascular adaptation, body fat/weight control, less bone loss caused by lactation, and less stress incontinence. Studies have generally indicated the importance of regular exercise in the postpartum period. Studies have generally indicated the importance of regular exercise in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

1. must be score of 13 and over in the Edinburgh Postpartum Depression Scale (EPDS),
2. must being between 19 and 40 years old,
3. must had a spontaneous vaginal delivery between the 38th and 42nd weeks of pregnancy,
4. must had a healthy newborn baby with 2500 gr and over

Exclusion Criteria:

1. postpartum obstetric complications
2. psychiatric disease history before or during pregnancy

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Effect of exercise | 4 week
  questionnaire and scale, Edinburgh Postpartum Depression Scale (EPDS) The screening scale, developed by Cox et al. (1987), aimed to identify depression risk in women in the postpartum period. It's a self-report scale that is composed of 10 items aiming to measure the individual's psychological state within the past 7 days. Each item is rated on a four-point Likert scale between 0 and 3 ("Yes, all the time", "Yes, most of the time", "No, not very often", and "No, not at all". Total score ranges between 0 and 30. Higher scores indicate the severity of depression. Aydin et al. (2004) performed the reliability and validity of the scale and identified the cut-off point for Turkish women as 12.5

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Şimşek Küçükkelepçe, Adi̇yaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No